CLINICAL TRIAL: NCT06357858
Title: Biomarker Driven Phase 1/1b Trial of ASTX727 and Nivolumab in Patients With Recurrent / Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: ASTX727 and Nivolumab in Squamous Cell Carcinoma of the Head and Neck
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE6323
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Head and Neck; Metastatic Squamous Cell Carcinoma; Head and Neck Squamous Cell Carcinoma
Keywords: ASTX727; Nivolumab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — decitabine and cedazuridine drug combination; Decitabine; cedazuridine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral Decitabine + Nivolumab (Experimental): Oral decitabine (ASTX727) will be administered during D1-5 (DL1) or D1-4 (DL1-1) followed by Nivolumab on D8 with every 4 week cycle. The expected minimum treatment cycle is 2 and maximum treatment cycle of 6. However, treatment can be continued until disease progression.
  Interventions: Drug: INQOVI (decitabine and cedazuridine); Drug: Nivolumab

INTERVENTIONS:
Drug: INQOVI (decitabine and cedazuridine) — Oral decitabine (ASTX727) will be administered during D1-5 (DL1) or D1-4 (DL1-1).
  Other Names: ASTX727
Drug: Nivolumab — Nivolumab will be administered on D8 with every 4 week cycle.
  Other Names: OPDIVO

SUMMARY:
The goal of this clinical trial is to see if the combination of experimental drug ASTX727 and Nivolumab enhances the antitumor immune response in participants will recurrent or metastatic squamous cell carcinoma of the head and neck.

Participants will take a pill called ASTX727 for 4 or 5 days every month followed by an injection of Nivolumab one week after the first dose of study medication.

DETAILED DESCRIPTION:
Anti PD1 inhibitor (Pembrolizumab, Nivolumab) is approved for recurrent/metastatic HNCC. However, response rates to Pembrolizumab or Nivolumab monotherapy are as low as 16-19%, underscoring the presence of immune evasion mechanisms. One of the main immune escape mechanisms described in HNSCC is poor tumor microenvironment characterized by defective HLA class I processing and antigen presentation, which allows tumor cells to evade their detection and destruction by cytotoxic CD8+ T-cells. Mutations or downregulation of the expression of HLA class I component including beta-2- microglobulin (β2M) and antigen processing machinery (APM) genes have been correlated with poor prognosis of HNSCC. Recent studies showed that de novo DNA methylation programs renders terminal T cell exhaustion and subsequent exhausted T cells are refractory to PD-1 blockade mediated rejuvenation. Pretreatment with DNA methyltransferases (DNMT) inhibitor prior to PD-L1 blockade showed enhancement of T cell responses and tumor control during PD-1 inhibitors in mice. A pilot study of novel combination of antiPD-1 and decitabine was conducted in patients with refractory or recurrent AML. The showed a best response of stable disease or better in 6 of 10 patients in patients with R-AML. A phase II clinical trial of anti-PD-1 camrelizumab plus decitabine, in relapsed/refractory Hodgkin lymphoma showed CR rate of 79% with decitabine plus camrelizumab compared to 32% with camrelizumab alone. Based on the promising results of decitabine enhances immune response and antitumor activity shown in both preclinical and preliminary clinical data from the phase II trial of hematological malignancies, I hypothesize that ASTX727 (oral decitabine and cedazuridine) changes DNA methylation status which may enhance the antitumor immune response by modulating tumor immune microenvironment and promoting increased tumor-infiltrating lymphocytes, which may enhance response to anti-PD1 inhibitor in R/M HNSCC patients

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed recurrent or metastatic HNSCC considered incurable by local therapies and eligible to receive anti-PD-L1 as first-line treatment (PD-L1 positive with combined positive score (CPS) ≥1 as evaluated in pre-screening).
* Participants must have primary tumor locations in following; oral cavity, hypopharynx, or larynx (nasopharynx is not allowed).
* Participants must have not received prior therapies for this disease, no systemic therapy administered in the recurrent or metastatic setting (except for systemic therapy completed within 6 months or > 6 months if given as part of multimodal treatment for locally advanced disease).
* Participants must have not received prior treatment with immune checkpoint inhibitors.
* Participants can provide archival tumor tissue not older than 12 months from a core or excisional biopsy for PD-L1 pre-screening using the PD-L1 IHC 22C3 pharmDx assay.
* Participants must have lesions amenable to obtain pre-treatment tumor biopsies in screening period after eligibility confirmation and before start of treatment and on- treatment tumor biopsies on C1D8 & C3D8 after start of treatment if lesions are still present at that time. If a recent archival biopsy is obtained within 3 months prior to start of treatment, this biopsy can be used as a pre-treatment biopsy.
* Participants should be age >18 years.
* Participants should have ECOG Performance status ≤ 2.
* Participants should have ability to swallow pills (participants will have to demonstrate the ability to swallow a placebo during screening).
* Participants must have normal organ and marrow function as defined below:

  * Hemoglobin ≥ 9.0 g/dl
  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelet count ≥ 100,000/mcL
  * Total bilirubin within normal institutional limits (Gilbert's syndrome related elevated bilirubin is accepted as long as levels have been stable within last 3 months).
  * AST (SGOT) ≤ 2.5 X institutional upper limit of normal
  * ALT (SGPT) ≤ 2.5 X institutional upper limit of normal
  * Serum Creatinine within normal institutional limits
* Women of child-bearing potential and sexually active men with female partners of child-bearing potential must agree to use a highly effective method of contraception beginning with the first dose of study therapy and for the duration of their participation in the study. This is expected for the entire duration of the study period through 6 months after the last dose. Highly effective methods of contraception include: female sterilization (tubal ligation, bilateral oophorectomy, and/or hysterectomy); male sterilization (at least 6 months prior to screening); intrauterine device; and oral, injected, or implanted hormonal contraception AND barrier methods of contraception. Women of child-bearing potential must have documented negative pregnancy test prior to start of investigational treatment regimen. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with progressive disease within six months of completion of curatively Intended systemic treatment for locoregionally advanced HNSCC.
* Participants with history of severe immune related adverse effects from prior immunotherapy, except hypothyroidism clinically stable on hormone replacement treatment and controlled type 1 diabetes. All other endocrinopathies are excluded even if controlled with medications.
* Participants with Grade ≥ 3 infections within 4 weeks before the first study drug administration. Clinically active infections > Grade 1 within 2 weeks before the first study drug administration.
* Participants with previous or active myocarditis/myositis in history (independent of cause).
* Participants with pneumonitis, idiopathic pulmonary fibrosis, organizing, interstitial lung disease active or history of autoimmune disease. . Autoimmune thyroid disease as well as other non-life threatening autoimmune diseases such as vitiligo or autoimmune alopecia that don't require systemic immunosuppression are not excluded.
* Participants with known human immunodeficiency virus (HIV) infection, uncontrolled active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
* Participants with treatment with systemic immunosuppressant medications within 2 weeks before the first study drug administration. However, low-dose steroid use (prednisone equivalent <=10mg daily) for other reasons is allowed.
* Participants receiving any other investigational agents.
* Participants with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants with confirmed COVID-19 within 7 days prior to start treatment will be excluded, however upon recovery with confirmation of negative COVID test, participant can be reconsidered for the study.
* Participants with a history of hypersensitivity to active or inactive excipients of ASTX727 or nivolumab or drugs with a similar chemical structure or class to either agent.
* Participants with any other condition which in the Investigator's opinion would not make the participant a good candidate for the clinical trial.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics Effect of ASTX727 on global DNA methylation status | 12 months after completion of treatment
  To find a biologically effective dose of ASTX727 in this clinical trial, levels of global DNA methylation at pre- versus post-ASTX727 will be compared using Wilcoxon signed-rank test.
Immunogenicity of ASTX27 in combination with Nivolumab | 12 months after completion of treatment
  To investigate the whether DNA methylation status affect immunologic biomarkers, changes in methylation status at pre-, post-ASTX727 and on treatment of ASTX727 plus Nivolumab will be correlated with the changes in immunologic biomarkers.
Maximum Tolerated Dose | 12 months after completion of treatment
  Establish the maximum tolerated dose (MTD) in Phase I part 1.
Safety of ASTX | 12 months after completion of treatment
  Assess safety of ASTX in combination with Nivolumab.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 12 months after completion of treatment
  The true objective response rate will be estimated based on the number of responses using a binomial distribution and its confidence interval will be estimated using Wilson's method.
Overall Survival (OS) | 12 months after completion of treatment
  Overall survival will be measured from the date of enrollment to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Kyunghee Burkitt, DO, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Compiled and analyzed patient data will be published upon study completion. Publisher may request Protocol and Statistical Analysis Plan.